CLINICAL TRIAL: NCT05552547
Title: Home BP Monitoring for Diagnosis of Hypertension in African American Adolescents
Brief Title: Home BP Monitoring
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Goutham Rao, MD, Chairman, Department of Family Medicine and Community Health, University Hospitals Cleveland Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY20221105
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: High Blood Pressure
Keywords: African American Teen; Home blood pressure monitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Blood Pressure Machine (Active Comparator): Participants will be asked to measure blood pressure twice daily for three days in a row.
  Interventions: Device: Home Blood Pressure Machine
- 24-Hour Blood Pressure Machine (Experimental): Participants will be asked to wear this machine for 24 hours.
  Interventions: Device: 24-Hour Blood Pressure Machine

INTERVENTIONS:
Device: Home Blood Pressure Machine — Participants will be asked to measure blood pressure twice daily for three days in a row at home.
  Arms: Home Blood Pressure Machine
Device: 24-Hour Blood Pressure Machine — Participants will be asked to wear the machine for 24 hours.
  Arms: 24-Hour Blood Pressure Machine

SUMMARY:
Most cases of high blood pressure in teens are missed for a number of reasons. One reason is that the most common way to make a diagnosis is to make three or more blood pressure measurements in a doctor's office on separate days. This can be inconvenient. Also, measuring blood pressure in the office might be inaccurate, since children (including teens) might have high values in the office but normal values at home. For these reasons, investigators wish to study a different way to identify teens with high blood pressure. Home BP measurements have been used in Europe to make a diagnosis, but not yet in the United States, and never in a higher risk population of teens. African American teens are at higher risk for high blood pressure than other teens. Investigators will compare the values received from the home BP machines to another method (24 hour ambulatory BP monitoring or ABPM) which is the best standard for diagnosis. Investigators also want to learn more about participants experience and their child's experience with both methods. A small sample of participating teens and parents will be invited to participate in short telephone interviews. This study plans to enroll a total of 750 teens at UH. Recruitment will not take place from other organizations.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify or identified by a parent as African-American or of partly African American ancestry

Exclusion Criteria:

* Prior hypertension diagnosis
* Prescribed BP medication
* History of congenital heart disease
* History of solid organ transplant
* Prescribed and using stimulants and other medications on a regular basis known to raise blood pressure such as testosterone and nicotine replacement

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 750 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who meet criteria for hypertension based on average home BP reading. | Up to 2 weeks
Number of participants who meet criteria for hypertension based on 24-hour ambulatory BP reading. | Up to 24 hours
Percent agreement between home BP-reading based diagnosis versus 24-hour ABPM | Up to 2 weeks
True positive rate -- Number of home bp positives over ABPM positives | Up to 2 weeks
True negative rate -- Number of home bp negatives over ABPM negatives | Up to 2 weeks

SECONDARY OUTCOMES:
Number of subjects who complete home BP protocol | Up to 2 weeks
Number of subjects who complete both home BP verus 24-hour ABPM protocols | Up to 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rao Goutham, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No